CLINICAL TRIAL: NCT04547400
Title: Relationship of Position Sense With Gait and Balance in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, Research Assistant, Gazi University
Other Study IDs: 2020-123
Record Dates: First submitted 2020-09-06; First posted 2020-09-14 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Gait; Balance; Sensation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Multiple Sclerosis: MS patients (EDSS: 0-5,5)
  Interventions: Other: assessment
- Healthy group: Healthy individuals without chronic disease
  Interventions: Other: assessment

INTERVENTIONS:
Other: assessment — Assessments of balance, gait, lower extremity position sense, and foot sole sense

SUMMARY:
Balance and gait disturbances are among the most common problems in patients with Multiple Sclerosis (MS). There is evidence of decreased foot sole sensation in MS patients. Studies conducted in healthy individuals have revealed the relationship between balance and foot sole sensation. These studies have demonstrated that sensory feedback from the cutaneous receptors of the foot sole plays an important role in maintaining balance. However, it is not yet known clearly to what extent the sensory impairment seen in MS patients affects balance and gait disorders.

The aim of this study is to examine the relationship between lower extremity position sense and foot sole sense with gait and balance in MS patients.

DETAILED DESCRIPTION:
Patients with MS between 0-5,5 score according to the Extended Disability Status Scale (EDSS) and healthy individuals of similar age and sex to patients will be included in the study. The balance, gait, lower extremity position sense, and foot sole sense will be evaluated.

The researchers will use t-tests to compare for quantitative variables and chi-square for the categorical variables between groups. In addition, the researchers will examine the correlations between balance, gait, lower extremity position sense, and foot sole using by Pearson bivariate correlations.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age Having a diagnosis of "Multiple Sclerosis" by a specialist physician Relapse free in the last 3 mounts Having an ambulatory status (Expanded Disability Status Scale score ≤ 6 ) No diagnosis of depression

Exclusion Criteria:

* Any cardiovascular, orthopedic, visual, hearing and perception problems that may affect the results of the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ambulatory sample
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Gait | 5 minutes
  Gait parameters will be assessed via the G-Walk on two separate occasions. The G-Walk is a device that is worn on the waist via an elastic belt. The G-Walk is built with a triaxial accelerometer 16 bit/axes with multiple sensitivity, a triaxial magnetometer 13 bit and a triaxial gyroscope 16 bit/axes with multiple sensitivity. This hardware is capable of acquiring and transmitting data to a computer through a Bluetooth connection and at the end of each analysis an automatic report containing the gait assessment results is ready to be analyzed.
  Gait symmetry values of the right and left sides are obtained within this report. While the symmetry index ranges from 0 to 100, a value closer to 100 indicates that the gait is more symmetrica
Balance | 10 minutes
  The Modified Sensory Organization Test, which is performed using computerized posturography, measures postural sway in response to 4 different sensory conditions is measured using a force platform.

SECONDARY OUTCOMES:
Light touch-pressure sensation | 10 minutes
  Light touch-pressure sensation will be assessed using a full Semmes-Weinstein Monofilament (SWM) test kit (North Coast Medical, San Jose, CA, USA).
Vibration sensation | 10 minutes
  Duration of vibration sensation will be measured using 128-Hz frequency tuning fork (Elcon1 Medical Instruments, Tuttlingen, Germany).
Two-point discrimination | 10 minutes
  Two-point discrimination sensation of the foot sole will be evaluated using an aesthesiometer (Baseline1, White Plains, New York, USA).
position sensation of knee joint | 5 minutes
  Open kinetic chain position of both knees will be evaluated using a Dualer IQ Digital Inclinometer (J-Tech Medical, Midvale, UT, USA).
Knee proprioception | 10 minutes
  Knee proprioception will be evaluated with the active joint reposition test using the isokinetic system (Cybex Norm, Humac, CA, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Cagla Ozkul, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cattaneo D, Jonsdottir J. Sensory impairments in quiet standing in subjects with multiple sclerosis. Mult Scler. 2009 Jan;15(1):59-67. doi: 10.1177/1352458508096874. Epub 2008 Oct 9. PMID 18845654
- [Background] Chung LH, Remelius JG, Van Emmerik RE, Kent-Braun JA. Leg power asymmetry and postural control in women with multiple sclerosis. Med Sci Sports Exerc. 2008 Oct;40(10):1717-24. doi: 10.1249/MSS.0b013e31817e32a3. PMID 18799980
- [Background] Eils E, Behrens S, Mers O, Thorwesten L, Volker K, Rosenbaum D. Reduced plantar sensation causes a cautious walking pattern. Gait Posture. 2004 Aug;20(1):54-60. doi: 10.1016/S0966-6362(03)00095-X. PMID 15196521
- [Background] Roll R, Kavounoudias A, Roll JP. Cutaneous afferents from human plantar sole contribute to body posture awareness. Neuroreport. 2002 Oct 28;13(15):1957-61. doi: 10.1097/00001756-200210280-00025. PMID 12395099